CLINICAL TRIAL: NCT03237949
Title: Comparative Effectiveness of Text Messaging and Telephone Counseling for Supporting Post-discharge Quit Attempts Among Hospitalized Smokers in Brazil
Brief Title: Text Messaging and Telephone Counseling for Supporting Post-discharge Quit Attempts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1.939.046
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Tobacco Use Cessation; Tobacco Use Disorder
Keywords: Tobacco Use Disorder; Hospitalized patients; Text message; Motivational Interview; Substance-Related Disorders; Behaviors and Mental Disorders
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use Disorder; Substance-Related Disorders; Behavior; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phone counseling (Active Comparator): The patient will receive standard care inside the hospital. After discharge the active comparator group will receive four phone counseling sessions. The sessions will provide basic information about smoking and successful quitting. The counselor will use motivational interview techniques to build coping skills with the goal of helping the participant build and implement a quit plan. The counseling timing, duration, and content will be consistent with guideline-based recommendations.
  Interventions: Behavioral: Phone counseling
- Text message (Experimental): The patient will receive standard care inside the hospital. After discharge the experimental group will receive extended care including text messages. Participants in this arm will be offered up to 30 text messages to help implement the quit plan discussed during the hospitalization. Patients motivated to quit in the next 30 days or that had already quit will receive 30 messages and patients unwilling to quit will receive 16 messages. The messages content follows the self efficacy theory.
  Interventions: Behavioral: Text message

INTERVENTIONS:
Behavioral: Phone counseling — Four telephone counseling sessions using a motivational interviewing approach
  Arms: Phone counseling
Behavioral: Text message — 30 messages (2 per day) and patients unwilling to quit 16 (2 per day). The messages follows the self efficacy theory. The messages follows the self efficacy theory.
  Arms: Text message

SUMMARY:
This is an extension of a previous feasibility study (Clinical Trials Registry - NCT02571244). The actual study is a research aimed to compare the effectiveness of telephone counseling and personalized text messages (TM) for supporting post-discharge quit attempts among hospitalized smokers, with focus on smoking cessation as the main outcome. Smokers patients will receive brief interventions and nicotine replacement therapy during the hospitalization. After discharge smoker patients will be allocated into a intervention or control arm. In the first and third months, after randomization, the patients will be contact to smoke abstinence assessment.

DETAILED DESCRIPTION:
This is an extension of a previous feasibility study (Clinical Trials Registry - NCT02571244). Background: Research suggests that smokers who receive treatment inside the hospital and post-discharge follow up for at least a month is most likely to quit smoking than those who didn't receive any intervention. The current challenge is to know the best way to support post-discharge quit attempts in the Brazilian context. Objective: The aim of this study is compare the effectiveness of personalized text messages (TM) and telephone counseling to support smoking cessation between post discharge patients. Methods: All patients admitted to the University Hospital of Juiz de Fora (HU/UFJF), between 06/2017 to 11/2018, will be asked about the cigarettes consumption in the last 30 days. Smokers patients will receive brief interventions and nicotine replacement therapy during hospitalization. After discharge these patients will be allocated into an intervention or control arm. The intervention group will receive mobile phone TM twice a day up to fifteen days. The control group will receive usual care (four telephone counseling sessions using motivational interviewing approach). Results: At the first and third months, after randomization, the patients will be contacted for smoke abstinence assessment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Smoked cigarettes in the last 30 days (even a puff)
* Have own mobile phone
* Have received at least one text message in the last year
* Have no problem with the mobile phone signal

Exclusion Criteria:

* Don't have a mobile phone
* Unstable cognitive or physical condition
* Physical or breath contact restrictions
* Intensive care units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Self Reported Smoking Abstinence | Smoking abstinence at the first month after randomization
  No smoking (even a puff) in the past 7 days at the first month follow up.

SECONDARY OUTCOMES:
Self Reported Smoking Abstinence | Smoking abstinence at the third month after randomization
  No smoking (even a puff) in the past 7 days at the third month after randomization.
Carbon monoxide verified Smoking Abstinence | At third-month follow up
  Carbon monoxide verified Smoking Abstinence at third-month follow up. Abstinence defined as Carbon monoxide ≤ 6.
Reduction of Daily Cigarettes Consumption From Baseline | At the third month after randomization
  The self reported daily cigarettes consumption at the third month after randomization will be compared to the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- University Federal Hospital of Juiz de Fora, Juiz de Fora, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] do Amaral LM, Ronzani TM, Cruvinel E, Richter K, Oliveira Andrade R, Lanzieri IO, de Macedo ACDAD, Leite ICG. Text messaging interventions to support smoking cessation among hospitalized patients in Brazil: a randomized comparative effectiveness clinical trial. BMC Res Notes. 2022 Mar 26;15(1):119. doi: 10.1186/s13104-022-06002-6. PMID 35346351
- Available data/document: Study Protocol: NCT02571244 — https://clinicaltrials.gov — This protocol is an extension of a previous research:Telephone Counseling and Text Messaging for Supporting Post-discharge Quit Attempts Among Hospitalized Smokers in Brazil, a feasibility study.